CLINICAL TRIAL: NCT06642506
Title: Oncometabolome and MALDI-MSI in Upper GI Carcinomas - Chemosensitivity in Esophageal Carcinoma.
Status: Active, not recruiting | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Max Planck Institute of Biochemistry, Department of Proteomics and Signal Transduction, MÃ¼nchen, Germany (Unknown); Dr. von Haunersches Children's Medical Hospital, University of Munich, Germany (Other)
Responsible Party: Principal Investigator, Ilja Balonov, MD, Principal Investigator, Ludwig-Maximilians - University of Munich
Other Study IDs: 24-0606
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Esophagus Adenocarcinoma; Esophagus Cancer; Metabolome; Mass Spectrometry; Precision Medicine; Oncology Patients Receiving Chemotherapy; Metabolomics; Chemoresistance
Keywords: Oncometabolome; Metabolomics; Mass Spectrometry Imaging; Esophagus Cancer; Chemosesitivity
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Tumortissue Adjacent normal tissue Blood Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Primary resection: Patients with esophageal adenocarcinoma who underwent esophagectomy without prior neoadjuvant therapy.
- Regression Grade 1: Patients with esophageal adenocarcinoma who received four cycles of neoadjuvant FLOT chemotherapy and subsequently underwent oncological esophagectomy. Final pathology revealed a regression grade of 1 according to the Becker classification.
- Regressions Grade 3: Patients with esophageal adenocarcinoma who received four cycles of neoadjuvant FLOT chemotherapy and subsequently underwent oncological esophagectomy. Final pathology revealed a regression grade of 3 according to the Becker classification.

SUMMARY:
Locally advanced adenocarcinoma of the esophagus is a leading cause of death from malignant disease in Germany and has been characterized on a molecular level in recent years. This retrospective observational study deals with patients after esophagectomy with different risk constellations of esophageal carcinoma. An early and individualized therapy of this tumor in an approach of precision oncology significantly improves the prognosis. The metabolomic profile plays a central role in tumor plasticity and oncological outcome. At the same time, these factors affect the efficacy of chemotherapy and need to be investigated in more detail at the molecular level. A central element of this study is the investigation of phospholipid metabolism locally in tumor tissue, in adjacent normal tissue in terms of the tumor microenvironment and systemically in blood plasma. The focus lies on the validation of known oncometabolites that significantly influence tumor sensitivity to chemotherapy.

By combining mass spectrometry imaging using matrix-assisted laser desorption ionization - mass spectrometry imaging (MALDI-MSI) with metabolomics using liquid chromatography tandem mass spectrometry (LC-MS/MS), the metabolic profile of tumors can be analyzed in detail, allowing conclusions to be drawn about chemo-insensitive and therapeutically challenging tumors. Both mass spectrometric methods are used to understand the heterogeneous metabolism of the tumors and to describe possible constellations that are associated with increasing chemoresistance. For precise investigation, the cohort under investigation is divided into two patient collectives. Patients with a regression grade 1 after four sessions of FLOT chemotherapy are compared with a regression grade 3 according to Becker in the postoperative pathological assessment. This facilitates the development of personalized therapeutic approaches tailored to the individual oncological profiles of the tumors. The study is complemented by conventional HE microscopic examinations of the tumor itself and the tumor microenvironment, which allow to analyze the morphology and its correlation with metabolic alterations in the tissue. We hypothesize that adenocarcinoma of the esophagus with regression grade 1 encompasses a fundamentally distinct metabolic profile than adenocarcinoma of the esophagus with regression grade 3. Consequently, a stratification parameter within the local tumor metabolism and the tumor microenvironment exists, which correlates with the systemic response to neoadjuvant chemotherapy in blood plasma.

The primary aim of the study is to create a comprehensive metabolic profile that clearly identifies tumors with a regression grade 1 versus a regression grade 3 according to Becker. This will be used to improve diagnostics and develop personalized treatment strategies that increase treatment efficiency and patients' chances of survival.

This is ultimately carried out with the intention of achieving an improved survival rate and a higher quality of life for patients with locally advanced esophageal cancer. The comprehensive analysis of the tumor microenvironment and the morphological and metabolic profiles should provide new insights into the mechanisms of tumor progression and resistance, which in turn will form the basis for future translational research and treatment approaches. The findings from this study have the potential to change the way esophageal cancer is treated by contributing to the development of stratified therapeutic approaches tailored to the molecular subtype of esophageal cancer.

DETAILED DESCRIPTION:
Introduction Esophageal cancer is one of the most common types of cancer worldwide. However, the incidence of esophageal cancer varies significantly by region, with higher rates observed in some countries such as Japan and South Korea. Tumors detected early have a better prognosis than advanced tumors. The 5-year survival rates for patients with esophageal cancer vary depending on the stage from 90% for localized tumours to only 5% in advanced stages (> T2, N+), whereby "patient" always refers to both genders. As the majority of patients are mainly diagnosed at a locally advanced stage, multimodal treatment is currently recommended in most cases before curative resection. The success of the systemic therapy, which in Germany is usually carried out as chemotherapy alone with the FLOT protocol or as radiochemotherapy with the CROSS protocol, is assessed postoperatively in the final histological evaluation by means of the degree of regression. According to Becker, the resulting degrees of regression are graded into stages 1 to 3, with grade 1 reflecting almost complete regression after systemic therapy and grade 3 indicating a postoperative residual tumor with > 50 % vital tumor cells and thus a poor response to neoadjuvant therapy.

The reason for favorable versus a poor response in esophageal adenocarcinoma cannot lie solely in the patients clinical characteristics and genetic subtype. Rather, the metabolic phenotype plays a decisive role. However, the metabolic phenotype of esophageal adenocarcinomas with different regression grade has not yet been sufficiently researched.

Rationale The oncological outcome of the esophageal adenocarcinoma depends on various factors, including in particular tumor size, tumor metabolism and the growth pattern of the primary tumor and infiltrated lymph nodes. An advanced tumor size is associated with an increased risk of local and systemic metastases and a poorer prognosis. At the same time, tumor size is associated with altered metabolic activity, particularly glycolysis. Tumor biology, which can be mapped using metabolomics, also plays an important role in the prognosis and treatment of these cancers. The expression of biomarkers such as HER2 and PD-L1 can also be of decisive importance both in the choice of therapy and in predicting the response to a particular treatment. However, locoregional growth, response to chemotherapy and tumor size also play a significant role in patient survival.

The tumor microenvironemt (TME), is frequently observed in esophageal carcinoma to induce cell proliferation and thus hardens the surrounding tissue and restricts blood flow to the tumor, which in turn reduces the effectiveness of chemotherapy and radiotherapy. Another key feature of tumor cell metabolism is the ability to extract nutrients from a frequently nutrient-poor microenvironment and use these nutrients to meet the demands of growth and proliferation. In this way, the TME gradually forms, encompassing cancer cells, the cytokine environment, the extracellular matrix, subgroups of fibroblasts and immune cells. Within this complex network of cancer cells and cancer-related metabolic products, the pro-tumorigenic environment plays a central role in stimulating tumor angiogenesis and promoting its invasiveness and metastatic potential. Certain tumor-associated metabolites are linked to aggressive cancer phenotypes, facilitated angiogenesis, promoted mutagenesis, and suppression of the immune system. However, the migration of cancer-related metabolites from the tumor itself and its microenvironment into the systemic bloodstream can be detected and quantified using state-of-the-art clinical mass spectrometry. Therefore, abnormal amino acid and phospholipid metabolism in various cancers plays a diverse and crucial role, and the potential impact of metabolic control and regulation within the tumor microenvironment is gaining increasing importance.

While metabolomics is already implemented in basic research, early detection, diagnosis, and therapy for metabolic diseases such as type 2 diabetes mellitus, there is currently a high demand for the application of targeted metabolomics in oncological diseases. In various entities, it has been observed that the metabolome within the TME harbors a significant alteration in amino acid and phospholipid metabolism. From a metabolic perspective, current investigations focus particularly on an increase in membrane-bound polar phospholipids and a decrease in apolar phospholipids and phosphate¬idylserines to characterize, for example, the response to chemotherapy.

In addition to this quantitative evaluation via targeted metabolomics of local metabolism in tumor tissue, the TME, and systemically in blood plasma, methods of mass spectrometry imaging allows for a qualitative assessment of tumor samples. Matrix-Assisted Laser Desorption/Ionization (MALDI) is a method for ionizing samples, where a matrix (usually a small organic acid) is mixed with the sample. The matrix-protein complex is then irradiated with a laser, leading to desorption and ionization of the molecules. In the case of esophageal carcinoma, MALDI-MSI is used to study tumor heterogeneity and visualize specific areas with high abundance of oncometabolites. The application of MALDI-MSI in other oncologic entities such as the pancreatic adenocarcinoma (PDAC) has provided specific insights into lipid metabolic changes associated with tumor growth and progression. For example, it has been found that certain lipids, such as phospholipids and sphingolipids, play a significant role in tumor biology. These changes in lipid metabolism can promote cancer cell proliferation and survival. These findings open new possibilities for the development of targeted therapies aimed at the altered lipid metabolism. For instance, areas of PDAC with higher proliferative and metabolic activity have been identified using glycerophosphocholine. Additionally, it was successfully observed that the glutamine/glutamate metabolism in tumor samples is significantly downregulated, indicating a fundamental reprogramming of cellular metabolism, which can be adequately represented using MALDI-MSI. Consequently, in blood and tissue samples from patients specifically diagnosed with esophageal carcinoma, functional histological examinations are conducted in addition to metabolomic studies to depict oncometabolites in tumor tissue and the tumor microenvironment.

The response to neoadjuvant therapy, in the era of approaches such as "NEOFLOTS," is more of a standard than a rarity, but to this day, no pre-therapeutic analysis for patient identification serves as its foundation. In terms of surgery in the locally advanced setting, which can lead significantly more patients to resection, this appears to be of great relevance. Current studies, particularly the correlation between the tumor's pattern of spread and its metabolism, show a clear association between these two characteristics and oncological outcome parameters. With sufficient knowledge of patient-specific tumor characteristics, it is possible to identify patients who, for example, would not benefit from systemic therapy due to their tumor metabolome, and should instead be directed to resection as quickly as possible.

Modern medicine inevitably follows a multimodal therapeutic approach. It is of great importance to individualize the final therapy decision as much as possible for each patient. This is only possible by considering all potential tumorigenic aspects. The underlying study aims to bridge the gap between newer approaches such as metabolism, and the pattern of tumor heterogeneity and spread. Up until now, the metabolomic properties of these tumors have barely been incorporated into diagnosis and therapy. Moreover, the TME in the upper gastrointestinal tract remains largely unexplored. However, studies in lung carcinoma have already shown changes in chemotherapy response depending on the TME. A joint investigation of the metabolome, cellular morphology in hematoxylin-eosin (HE) histological sections, and molecular constellation using MALDI-MSI, as well as an investigation of correlations between these two aspects, has not yet been conducted in esophageal carcinoma.

Hypothesis We hypothesize that (I) adenocarcinoma of the esophagus with regression grade 1 encompasses a fundamentally distinct metabolic profile than adenocarcinoma of the esophagus with regression grade 3. (II) Consequently, a stratification parameter within the local tumor metabolism and the tumor microenvironment exists, which correlates with the systemic response to neoadjuvant chemotherapy in blood plasma.

Objectives Primary objective The primary objective is to evaluate phospholipids in three compartments as a new stratification parameter for patients with adenocarcinoma of the esophagus with different responses to chemotherapy after four cycles of neoadjuvant FLOT chemotherapy, followed by surgery for locally advanced esophageal cancer.

Primary endpoint The primary endpoint for beneficial response to neoadjuvant chemotherapy is defined by the regressions grad according to Becker. The primary endpoint for phospholipids as a new parameter for response to chemotherapy is the increase of phosphatidylcholines in the local tumor tissue in the adjacent normal tissue and in blood samples.

Secondary objectives To determine a metabolic profile which shows a significant correlation between patients with regression grade 1 after neoadjuvant chemotherapy compared to regression grade 3.

To evaluate the expression and distribution of the identified oncometabolites in tumor tissue and adjacent tissue.

Secondary endpoints The metabolic profile will be carried out by LC-MS/MS, following multivariate analysis The expression and distribution of oncometabolites will be evaluated by MALDI - MSI

Study design This is a retrospective, observative, open label study of the correlation between phospholipid metabolism and the regressions grade in study participants with locally advanced esophageal cancer after four cycles of neoadjuvant chemotherapy according to the FLOT protocol.

Approximately 20 study participants with newly diagnosed adenocarcinoma of the esophagus with a tumor stage of uT2, uN+, cM0 or uT3, cNx, cM0 will be first treated with FLOT, following open or minimal-invasive esophagectomy. Baseline medical imaging with CT/MRI, according to standard clinical practice, is performed within 28 days before neoadjuvant treatment start. First tumor assessment after neoadjuvant treatment with CT scan/MRI is scheduled within two weeks before surgery. A second tumor assessment is planned within two weeks before adjuvant treatment start. Thereafter, every 12 weeks (+/- 2 weeks) up to end of treatment visit. In the period of follow up a CT/MRI will be performed every 12 weeks (+/- 2 weeks) for a time of 24 months.

Study population The study population consists of patients who underwent surgery for stomach or esophageal tumors between January 1, 2018, and January 31, 2024, at the Department of General, Visceral, and Transplantation Surgery. One prerequisite is the availability of fresh-frozen tumor tissue in the archive of the Department of General, Visceral, and Transplantation Surgery, as well as fresh-frozen tumor tissue from the institution's biobank (sample material request has been approved), and a complete clinical dataset with a five-year follow-up for each patient. The final cohort consists of patients for whom both the frozen biobank specimen, potentially with a serum sample, and the paraffin-embedded tumor tissue are available.

Flow-Chart and Events Schedule A study design has been established for the conduct of the investigation. The chromatographic, mass spectrometric, and immunohistochemical methods employed have already been validated, and compliance with Good Clinical Practice (GCP) regarding data management is ensured through appropriate standard operating procedures (SOPs). Since this is a retrospective data collection, the samples have already been stored in the in-house biobank at -80°C at the time of the application. Basic patient data are already stored in existing databases at our institution. All patients underwent surgery in the Clinic and Polyclinic for General, Visceral, and Transplant Surgery at the LMU Munich Hospital and were informed through the register of the Study, Documentation, and Quality Center (StuDoQ) of the German Society for General and Visceral Surgery (DGAV). The sample collection has already been conducted by the in-house biobank. Our patients have already consented to the collection and scientific utilization of samples during the initial sampling perioperatively. Upon retrieval, these samples are pre-processed in the laboratory for experimental surgery in preparation for metabolomic measurements. The pre-processing includes the careful thawing of the samples over a period of 24 hours, as well as the aliquoting of the samples in the surgical laboratory. Subsequently, the samples are transported to the location of the in-house MS core facility until measurement.

Clinical characteristics At baseline, a medical history have been obtained. The baseline examinations include weight (to be measured at the study site), height, ECOG Performance Status, measured blood pressure (BP), heart rate (HR), temperature and oxygen saturation by pulse oximetry at rest within 28 days prior to first cycle of neoadjuvant FLOT chemotherapy. Baseline signs and symptoms are those that are assessed within 14 days prior to first dose. Concomitant medication were collected from within 14 days prior to first cycle.

Baseline local laboratory assessments have been done within 14 days prior to first cycle and include: complete blood count with differential, liver function test (ALT, AST, total bilirubin and AP), serum urea level, uric acid, creatinine with creatinine clearance, phosphate, glucose, serum albumin, C-reactive protein, amylase, lipase, TSH, free T3 and free T4, tumor marker CEA and CA 19-9. Physical examinations, on study weight, ECOG performance status, vital signs and oxygen saturation have been assessed prior to neoadjuvant chemotherapy. Additional measures, including non-study required laboratory tests, should be performed as clinically indicated or to comply with local regulations. Additional testing or assessments may be performed as clinically necessary or where required by institutional or local regulations.

Screening or baseline assessments are to be performed within 28 days prior to treatment start. External CT scans/MRI performed before enrolment in the trial is feasible as baseline scan if performed no longer than 28 prior to first dose of study drug administration. In addition to the neck, chest, abdomen and pelvis all known sites of disease should be assessed at baseline. Subsequent assessments should include neck, chest, abdomen using the same imaging method and technique as used at baseline. Disease assessment with contrast-enhanced computed tomography (CT) scans acquired on dedicated CT equipment is preferred for this study. Conventional CT with IV contrast and MRI gadolinium should be performed with contiguous cuts of 10 mm or less slice thickness. Spiral CT should be performed using a 3- or 5-mm contiguous reconstruction. Should study participant have contraindication for CT MRI may be performed. In cases, application of CT IV contrast is contra-indicated ; tumor assessment should preferably be performed using a non-contrast CT scan of the chest and a contrast-enhanced MRI of the neck and abdomen.

Tumor measurements should be made by the same investigator or radiologist for each assessment whenever possible. Change in tumor measurements and tumor response will be assessed by the Investigator using the RECIST 1.1 criteria. Bone scan, PET scan and ultrasound is not adequate for assessment of RECIST 1.1 response in target lesions. Complementary CT and/or MRI or biopsy must be performed in such cases.

Doubtful, cutaneous, subcutaneous or lymph node lesions that are suspected should be confirmed by biopsy. Histological or cytological evidence of recurrence should be attempted in all cases except for brain metastases when safe and clinically feasible. An example when obtaining a biopsy to confirm recurrence may not be safe and clinically feasible is brain metastases.

Biomarker Assessment As the neoadjuvant setting offers the unique opportunity to achieve large tumor samples from patients after multimodal treatment, the study includes a comprehensive analysis of immune responses to private and shared antigens. These analyses rely on standardized collection of tissue and blood samples, which allow the planned metabolomic, massspectromeric and functional immunologic analyses.

Unfixed tumor specimens will be taken to our Institute of Pathology immediately following resection. Tumor tissue and normal tissue will be processed according to local diagnostic standards of procedure. In case of sufficient material, biopsies of tumor and normal tissue can be taken and stored in liquid nitrogen. As determined by the pathologist, additional fresh tumor tissue, which is not needed for pathological staging, will be transferred to the biobank. These samples will be analyzed by immunohistochemistry and molecular analyses, respectively.

Blood (45mL EDTA), plasma (20mL) and serum (4.5mL) samples have been obtained at screening and have been immediately transferred to the biobank.

Targeted metabolomics The LC-MS/MS method was validated based on the current guidelines for bioanalytical method validation from the European Medicines Agency (2011) and the U.S. Food and Drug Administration (2018). For LC-MS/MS measurements, an Agilent 1290 HPLC coupled with a QTRAP 6500+ MS system is used. Data acquisition and quantification are performed using Analyst 1.6.3. The analytical column is an Acquity UPLC Premier HSS T3 1.8 μm 2.1x50mm, and offline solid-phase extraction (SPE) is carried out using SepPak tC18 100 mg 96-well plates. Methanol and water of MS grade are obtained from VWR International GmbH. Formic acid, ammonium acetate, and acetic acid are sourced from Thermo Fisher Scientific Inc.. The extracted metabolites are eluted into a collection plate in two consecutive steps with 2 × 300 μl of methanol. After complete solvent evaporation at 50°C under a gentle nitrogen stream, the samples are reconstituted in 150 μl of methanol and diluted with 150 μl of water. A 10 μl aliquot of the extracted sample is injected into the HPLC system. Samples with concentrations exceeding the upper limit of quantification are reanalyzed after incubation. Each analysis run is preceded by a one-minute automatic re-equilibration. For each analyte, a quantifier and a qualifier transition are identified and optimized for maximum intensity. Isobaric compounds are baseline-separated from the analyte peaks.

The Biocrates MxP® Quant 500 XL Kit (Biocrates Life Sciences AG, Innsbruck, Austria) is used for the measurements, allowing the quantification of 106 small molecules in chromatography mode and 524 lipids in flow injection mode (FIA-MS/MS), thereby covering the major metabolic pathways. The kit includes a patented 96-well filter plate with pre-set internal standards, calibration standards, and quality controls, as well as a test sample for system suitability testing. The qualitatively and quantitatively obtained metabolites are exported as an Excel file and further processed in the surgical laboratory.

Mass spectrometry imaging The tumor tissue and adjacent normal tissue samples are dissolved in a matrix and applied to a MALDI plate. The samples are irradiated with a UV laser, causing the molecules to become ionized. The ionized molecules are then accelerated in an electric field, and their flight time is measured to determine the m/z ratio. Imaging experiments are performed using a rapifleX MALDI Tissuetyper MALDI-TOF/TOF mass spectrometer (Bruker Daltonik GmbH), equipped with a SmartBeam 3G laser. Tissues are measured in positive reflector mode with a spatial resolution of 25 μm and a mass range of 600-3,200 Da. Each measurement is externally precalibrated using a commercial peptide calibration mixture on the same target as the tissues at multiple positions. Tissues from all patients are measured on the rapifleX with a sampling rate of 1.25 GS/s and a pulsed ion extraction of 160 ns. After the MALDI-MSI measurements, the HCCA matrix is removed by washing the slide in 70% ethanol, followed by H&E counterstaining. High-resolution images of the stained sections were acquired using the Mirax Scan system (Carl Zeiss MicroImaging) and co-registered with the MALDI-IMS data for histological correlation.

Data Protection The provisions of data protection legislation will be observed. It is assured by the sponsor that all investigational materials and data will be irreversibly anonymized in accordance with data protection legislation before scientific processing. Trial study participants will be informed that their anonymized data will be passed on in accordance with provisions for documentation and notification pursuant to §12 and §13 of the GCP Regulations to the recipients described there. Study participants who do not agree that information may be passed on in this way will not be enrolled into the trial.

ELIGIBILITY:
Inclusion Criteria:

* Signed Written Informed Consent
* Study participants must have signed and dated an IEC approved written informed consent form in accordance with regulatory and institutional guidelines.
* Study participants must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests and other requirements of the study.
* Histologically confirmed, resectable adenocarcinoma of the esophagus (uT2, uN+, cM0 or uT3, cNx, cM0), with the following specifications:
* Medical and technical operability
* No preceding cytotoxic or targeted therapy
* No prior partial or complete tumor resection
* Male or female patients > 18 years of age at time of study entry
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Life expectancy of at least 12 months
* Adequate normal organ function as defined below. Screening laboratory values must meet the following criteria and should be obtained within 28 days prior to registration
* WBC ≥ 1500/μL
* Neutrophils ≥ 1000/μL
* Platelets ≥ 75 x103/μL
* Hemoglobin > 9.0 g/dL
* Serum creatinine ≤ 1.5 x institutional ULN or calculated creatinine clearance ≥ 40 mL/min (Cockcroft-Gault)
* AST/ALT ≤ 2,5 x institutional ULN
* Total Bilirubin ≤ 1.5 x institutional ULN
* Body weight > 30kg
* Reproductive Status
* Women of childbearing potential must have a negative serum or urine pregnancy test within one until two weeks prior to the start of neoadjuvant treatment and after surgery before starting adjuvant treatment.
* Women ≥ 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago.
* Women must not be breastfeeding.
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year.

Exclusion Criteria:

* Study participants with squamous cell carcinoma of the esophagus
* Prior treatment with chemotherapy, targeted therapy or radiotherapy for treatment of advanced cancer disease less than 5 years.
* Enrollment is possible for patients with:
* Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
* Adequately treated carcinoma in situ without evidence of disease
* Any other serious or uncontrolled medical disorder, active infections, physical exam findings, laboratory finding, altered mental status, or psychiatric condition that, in the opinion of the investigator, would limit a study participant's ability to comply with the study requirements, substantially increase risk to the study participant, or impact the interpretability or study results
* Active or prior documented autoimmune or inflammatory disorders. The following are exceptions to this criterion:
* Patients with vitiligo or alopecia
* Patients with hypothyroidism stable on hormone replacement
* Any chronic skin condition that does not require systemic therapy
* Patients with celiac disease controlled by diet alone.
* Inhaled or topical steroids and adrenal replacement steroid doses >10mg daily prednisone equivalent are permitted in the absence of active autoimmune disease.
* History of active primary immunodeficiency
* History of any allogenic organ transplantation with currently intake of immune suppressive treatment
* Patients with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity. FEV 1 < 75%
* Patients has known current symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. ∙
* Prisoners or study participants who are involuntarily incarcerated

Pregnancy or breastfeeding females

∙ Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy or 180 days after the last dose of durvalumab + tremelimumab combination therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with histologically confirmed esophageal adenocarcinoma who may be eligible for primary resection or neoadjuvant chemotherapy with four cycles of FLOT followed by esophagectomy, following discussion in the interdisciplinary tumor board.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-10-06 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Oncometabolome | From enrollment to the end of treatment at 10 weeks
  The primary endpoint is the metabolome of the tumor tissue, with a particular focus on significant differences in the composition of membrane lipids, amino acids, and carbohydrates between the group "Regressions Grade 1" and "Regressions Grade 3"

SECONDARY OUTCOMES:
Mass spectrometry imaging of the metabolome | From enrollment to the end of treatment at 10 weeks
  The expression and distribution of identified oncometabolites will be evaluated by MALDI - MSI

CONTACTS AND LOCATIONS:
Overall Officials: Ilja Balonov, Dr. med., Principal Investigator — Department of General, Visceral, and Transplant Surgery, Ludwig-Maximilians-University Munich, Germany; Jens Werner, Prof. Dr. med., Study Chair — Department of General, Visceral, and Transplant Surgery, Ludwig-Maximilians-University Munich, Germany
Locations (1):
- Department of General, Visceral and Transplantation Surgery, LMU University Hospital, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
Irreversibly anonymized data

REFERENCES:
- [Background] Schmidt HM, Gisbertz SS, Moons J, Rouvelas I, Kauppi J, Brown A, Asti E, Luyer M, Lagarde SM, Berlth F, Philippron A, Bruns C, Holscher A, Schneider PM, Raptis DA, van Berge Henegouwen MI, Nafteux P, Nilsson M, Rasanen J, Palazzo F, Rosato E, Mercer S, Bonavina L, Nieuwenhuijzen G, Wijnhoven BPL, Schroder W, Pattyn P, Grimminger PP, Gutschow CA. Defining Benchmarks for Transthoracic Esophagectomy: A Multicenter Analysis of Total Minimally Invasive Esophagectomy in Low Risk Patients. Ann Surg. 2017 Nov;266(5):814-821. doi: 10.1097/SLA.0000000000002445. PMID 28796646
- [Background] Low DE, Kuppusamy MK, Alderson D, Cecconello I, Chang AC, Darling G, Davies A, D'Journo XB, Gisbertz SS, Griffin SM, Hardwick R, Hoelscher A, Hofstetter W, Jobe B, Kitagawa Y, Law S, Mariette C, Maynard N, Morse CR, Nafteux P, Pera M, Pramesh CS, Puig S, Reynolds JV, Schroeder W, Smithers M, Wijnhoven BPL. Benchmarking Complications Associated with Esophagectomy. Ann Surg. 2019 Feb;269(2):291-298. doi: 10.1097/SLA.0000000000002611. PMID 29206677
- [Background] Kudo T, Hamamoto Y, Kato K, Ura T, Kojima T, Tsushima T, Hironaka S, Hara H, Satoh T, Iwasa S, Muro K, Yasui H, Minashi K, Yamaguchi K, Ohtsu A, Doki Y, Kitagawa Y. Nivolumab treatment for oesophageal squamous-cell carcinoma: an open-label, multicentre, phase 2 trial. Lancet Oncol. 2017 May;18(5):631-639. doi: 10.1016/S1470-2045(17)30181-X. Epub 2017 Mar 15. PMID 28314688
- [Background] Hingorani M, Goody R, Bozas G, Zahid K, Mitton DJ, Jain P, Wong V, Roy R. Neoadjuvant Management of Adenocarcinoma of the Esophagus and Esophagogastric Junction: Review of Randomized Evidence and Definition of Optimum Treatment Algorithm. Oncology. 2023;101(9):553-564. doi: 10.1159/000527716. Epub 2023 Apr 4. PMID 37015204
- [Background] Lombardi PM, Pansa A, Basato S, Giorgi L, Perano V, Marano S, Castoro C. Facing adenocarcinoma of distal esophagus and esophagogastric junction: a CROSS versus FLOT propensity score-matched analysis of oncological outcomes in a high-volume institution. Updates Surg. 2023 Jun;75(4):921-930. doi: 10.1007/s13304-023-01497-5. Epub 2023 Mar 29. PMID 36991302
- [Background] Gotze TO, Piso P, Lorenzen S, Bankstahl US, Pauligk C, Elshafei M, Amato G, Reim D, Bechstein WO, Konigsrainer A, Monig SP, Rau B, Schwarzbach M, Al-Batran SE. Preventive HIPEC in combination with perioperative FLOT versus FLOT alone for resectable diffuse type gastric and gastroesophageal junction type II/III adenocarcinoma - the phase III "PREVENT"- (FLOT9) trial of the AIO /CAOGI /ACO. BMC Cancer. 2021 Oct 29;21(1):1158. doi: 10.1186/s12885-021-08872-8. PMID 34715810
- [Background] Lorenzen S, Pauligk C, Homann N, Schmalenberg H, Jager E, Al-Batran SE. Feasibility of perioperative chemotherapy with infusional 5-FU, leucovorin, and oxaliplatin with (FLOT) or without (FLO) docetaxel in elderly patients with locally advanced esophagogastric cancer. Br J Cancer. 2013 Feb 19;108(3):519-26. doi: 10.1038/bjc.2012.588. Epub 2013 Jan 15. PMID 23322206
- [Background] Alexandrov LB, Nik-Zainal S, Wedge DC, Aparicio SA, Behjati S, Biankin AV, Bignell GR, Bolli N, Borg A, Borresen-Dale AL, Boyault S, Burkhardt B, Butler AP, Caldas C, Davies HR, Desmedt C, Eils R, Eyfjord JE, Foekens JA, Greaves M, Hosoda F, Hutter B, Ilicic T, Imbeaud S, Imielinski M, Jager N, Jones DT, Jones D, Knappskog S, Kool M, Lakhani SR, Lopez-Otin C, Martin S, Munshi NC, Nakamura H, Northcott PA, Pajic M, Papaemmanuil E, Paradiso A, Pearson JV, Puente XS, Raine K, Ramakrishna M, Richardson AL, Richter J, Rosenstiel P, Schlesner M, Schumacher TN, Span PN, Teague JW, Totoki Y, Tutt AN, Valdes-Mas R, van Buuren MM, van 't Veer L, Vincent-Salomon A, Waddell N, Yates LR; Australian Pancreatic Cancer Genome Initiative; ICGC Breast Cancer Consortium; ICGC MMML-Seq Consortium; ICGC PedBrain; Zucman-Rossi J, Futreal PA, McDermott U, Lichter P, Meyerson M, Grimmond SM, Siebert R, Campo E, Shibata T, Pfister SM, Campbell PJ, Stratton MR. Signatures of mutational processes in human cancer. Nature. 2013 Aug 22;500(7463):415-21. doi: 10.1038/nature12477. Epub 2013 Aug 14. PMID 23945592
- [Background] Kunzke T, Balluff B, Feuchtinger A, Buck A, Langer R, Luber B, Lordick F, Zitzelsberger H, Aichler M, Walch A. Native glycan fragments detected by MALDI-FT-ICR mass spectrometry imaging impact gastric cancer biology and patient outcome. Oncotarget. 2017 Jul 10;8(40):68012-68025. doi: 10.18632/oncotarget.19137. eCollection 2017 Sep 15. PMID 28978092
- [Background] Gaye MM, Ding T, Shion H, Hussein A, Hu Y, Zhou S, Hammoud ZT, Lavine BK, Mechref Y, Gebler JC, Clemmer DE. Delineation of disease phenotypes associated with esophageal adenocarcinoma by MALDI-IMS-MS analysis of serum N-linked glycans. Analyst. 2017 May 2;142(9):1525-1535. doi: 10.1039/c6an02697d. PMID 28367546
- [Background] Erich K, Reinle K, Muller T, Munteanu B, Sammour DA, Hinsenkamp I, Gutting T, Burgermeister E, Findeisen P, Ebert MP, Krijgsveld J, Hopf C. Spatial Distribution of Endogenous Tissue Protease Activity in Gastric Carcinoma Mapped by MALDI Mass Spectrometry Imaging. Mol Cell Proteomics. 2019 Jan;18(1):151-161. doi: 10.1074/mcp.RA118.000980. Epub 2018 Oct 7. PMID 30293968
- [Background] Streitz JM Jr, Madden MT, Marimanikkuppam SS, Krick TP, Salo WL, Aufderheide AC. Analysis of protein expression patterns in Barrett's esophagus using MALDI mass spectrometry, in search of malignancy biomarkers. Dis Esophagus. 2005;18(3):170-6. doi: 10.1111/j.1442-2050.2005.00488.x. PMID 16045579
- [Background] Balluff B, Rauser S, Ebert MP, Siveke JT, Hofler H, Walch A. Direct molecular tissue analysis by MALDI imaging mass spectrometry in the field of gastrointestinal disease. Gastroenterology. 2012 Sep;143(3):544-549.e2. doi: 10.1053/j.gastro.2012.07.022. Epub 2012 Jul 20. No abstract available. PMID 22820311
- [Background] Wang Y, Chen W, Li K, Wu G, Zhang W, Ma P, Feng S. Tissue-based metabolomics reveals metabolic signatures and major metabolic pathways of gastric cancer with help of transcriptomic data from TCGA. Biosci Rep. 2021 Oct 29;41(10):BSR20211476. doi: 10.1042/BSR20211476. PMID 34549263
- [Background] Hatogai K, Kitano S, Fujii S, Kojima T, Daiko H, Nomura S, Yoshino T, Ohtsu A, Takiguchi Y, Doi T, Ochiai A. Comprehensive immunohistochemical analysis of tumor microenvironment immune status in esophageal squamous cell carcinoma. Oncotarget. 2016 Jul 26;7(30):47252-47264. doi: 10.18632/oncotarget.10055. PMID 27322149
- [Background] Pun C, Luu S, Swallow C, Kirsch R, Conner JR. Prognostic Significance of Tumour Budding and Desmoplastic Reaction in Intestinal-Type Gastric Adenocarcinoma. Int J Surg Pathol. 2023 Sep;31(6):957-966. doi: 10.1177/10668969221105617. Epub 2022 Jun 20. PMID 35726174
- [Background] Liu J, Zhong L, Deng D, Zhang Y, Yuan Q, Shang D. The combined signatures of the tumour microenvironment and nucleotide metabolism-related genes provide a prognostic and therapeutic biomarker for gastric cancer. Sci Rep. 2023 Apr 24;13(1):6622. doi: 10.1038/s41598-023-33213-z. PMID 37095256
- [Background] Meier A, Nekolla K, Hewitt LC, Earle S, Yoshikawa T, Oshima T, Miyagi Y, Huss R, Schmidt G, Grabsch HI. Hypothesis-free deep survival learning applied to the tumour microenvironment in gastric cancer. J Pathol Clin Res. 2020 Oct;6(4):273-282. doi: 10.1002/cjp2.170. Epub 2020 Jun 27. PMID 32592447
- [Background] Dickerson LK, Carter JA, Kohli K, Pillarisetty VG. Emerging interleukin targets in the tumour microenvironment: implications for the treatment of gastrointestinal tumours. Gut. 2023 Aug;72(8):1592-1606. doi: 10.1136/gutjnl-2023-329650. Epub 2023 May 31. PMID 37258094
- [Background] Pardoll DM. Immunology beats cancer: a blueprint for successful translation. Nat Immunol. 2012 Dec;13(12):1129-32. doi: 10.1038/ni.2392. PMID 23160205
- [Background] King R, Hayes C, Donohoe CL, Dunne MR, Davern M, Donlon NE. Hypoxia and its impact on the tumour microenvironment of gastroesophageal cancers. World J Gastrointest Oncol. 2021 May 15;13(5):312-331. doi: 10.4251/wjgo.v13.i5.312. PMID 34040696
- [Background] Li W, Ng JM, Wong CC, Ng EKW, Yu J. Molecular alterations of cancer cell and tumour microenvironment in metastatic gastric cancer. Oncogene. 2018 Sep;37(36):4903-4920. doi: 10.1038/s41388-018-0341-x. Epub 2018 May 23. PMID 29795331
- [Background] Peng X, Chen Z, Farshidfar F, Xu X, Lorenzi PL, Wang Y, Cheng F, Tan L, Mojumdar K, Du D, Ge Z, Li J, Thomas GV, Birsoy K, Liu L, Zhang H, Zhao Z, Marchand C, Weinstein JN; Cancer Genome Atlas Research Network; Bathe OF, Liang H. Molecular Characterization and Clinical Relevance of Metabolic Expression Subtypes in Human Cancers. Cell Rep. 2018 Apr 3;23(1):255-269.e4. doi: 10.1016/j.celrep.2018.03.077. PMID 29617665
- [Background] Derks S, Nason KS, Liao X, Stachler MD, Liu KX, Liu JB, Sicinska E, Goldberg MS, Freeman GJ, Rodig SJ, Davison JM, Bass AJ. Epithelial PD-L2 Expression Marks Barrett's Esophagus and Esophageal Adenocarcinoma. Cancer Immunol Res. 2015 Oct;3(10):1123-1129. doi: 10.1158/2326-6066.CIR-15-0046. Epub 2015 Jun 16. PMID 26081225
- [Background] Zhang J, Bowers J, Liu L, Wei S, Gowda GA, Hammoud Z, Raftery D. Esophageal cancer metabolite biomarkers detected by LC-MS and NMR methods. PLoS One. 2012;7(1):e30181. doi: 10.1371/journal.pone.0030181. Epub 2012 Jan 23. PMID 22291914
- [Background] Schmidt DR, Patel R, Kirsch DG, Lewis CA, Vander Heiden MG, Locasale JW. Metabolomics in cancer research and emerging applications in clinical oncology. CA Cancer J Clin. 2021 Jul;71(4):333-358. doi: 10.3322/caac.21670. Epub 2021 May 13. PMID 33982817
- [Background] Otsuka R, Hayano K, Hayashi H, Uesato M, Murakami K, Toyozumi T, Matsumoto Y, Kurata Y, Nakano A, Matsubara H. ypTNM staging is a potentially useful prognostic stratification tool in patients with advanced gastric cancer after preoperative chemotherapy. Langenbecks Arch Surg. 2023 Mar 31;408(1):133. doi: 10.1007/s00423-023-02872-x. PMID 37000278
- [Background] Wang Z, Goodman M, Saba N, El-Rayes BF. Incidence and prognosis of gastroesophageal cancer in rural, urban, and metropolitan areas of the United States. Cancer. 2013 Nov 15;119(22):4020-7. doi: 10.1002/cncr.28313. Epub 2013 Aug 20. PMID 23963864